CLINICAL TRIAL: NCT07148414
Title: Phase 2 Study to Assess the Efficacy and Safety of SPY002-072 in Adults With Moderately to Severely Active Rheumatologic Disease
Brief Title: A Study of SPY072 in Rheumatic Disease
Acronym: SKYWAY-RD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spyre Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPY002-072-201
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Axial Spondyloarthritis; Rheumatic Diseases; Rheumatic Joint Disease; PsA (Psoriatic Arthritis); AxSpA; Rheumatologic Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Axial Spondyloarthritis; Rheumatic Diseases; Collagen Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Rheumatoid Arthritis, Dose Regimen 1 (Experimental): Participants will receive double-blind dosing regimen 1 of SPY072
  Interventions: Drug: SPY002-072
- Rheumatoid Arthritis, Dose Regimen 2 (Experimental): Participants will receive double-blind dosing regimen 2 of SPY072
  Interventions: Drug: SPY002-072
- Psoriatic Arthritis (Experimental): Participants will receive double-blind dose of SPY072
  Interventions: Drug: SPY002-072
- Axial Spondyloarthritis (Experimental): Participants will receive double-blind dose of SPY072
  Interventions: Drug: SPY002-072
- Rhematoid Arthritis Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo
- Psoriatic Arthritis Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo
- Axial Spondyloarthritis Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPY002-072 — Experimental
  Other Names: SPY072
  Arms: Axial Spondyloarthritis; Psoriatic Arthritis; Rheumatoid Arthritis, Dose Regimen 1; Rheumatoid Arthritis, Dose Regimen 2
Drug: Placebo — Matching Placebo
  Arms: Axial Spondyloarthritis Placebo; Psoriatic Arthritis Placebo; Rhematoid Arthritis Placebo

SUMMARY:
This is a multi-center, double-blind, placebo-controlled, Phase 2, proof-of-concept basket study with the goal of assessing the efficacy and safety of SPY072 compared to placebo in adults (aged ≥18 years) with rheumatic disease (RD).

DETAILED DESCRIPTION:
The basket study comprises of substudies in rheumatoid arthritis (RA), axial spondyloarthritis (axSpA) and psoriatric arthritis (PsA) as follows:

* RA substudy: Moderately to severely active RA despite treatment with conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs), biologic disease modifying anti-rheumatic drugs (bDMARDs), or targeted synthetic disease-modifying anti-rheumatic drugs (tsDMARDs)
* axSpA substudy: Moderately to severely active axSpA despite treatment with non-steroidal anti-inflammatory drugs (NSAIDS), bDMARDs, or tsDMARDs
* PsA substudy: Moderately to severely active PsA despite treatment with NSAIDs, csDMARDs, bDMARDs, or tsDMARDs

ELIGIBILITY:
Inclusion Criteria:

For rheumatoid arthritis:

* Moderate-to-severely active RA as defined by the presence of ≥4 swollen joints (based on 28 joint count) and ≥4 tender joints (based on 28 joint count) at Screening and Day 1.
* Documentation of ≥1 of the following:

  1. Positive test results for rheumatoid factor or anti-citrullinated peptide antibodies at Screening, OR
  2. Radiology report documenting bony erosions in hands or feet consistent with RA on previous radiographs
* Inadequate response (defined as signs and symptoms of persistently active disease, loss of response, or intolerance) to:

  1. ≥1 csDMARD treatment; AND/OR
  2. ≤2 classes of bDMARD/tsDMARD treatment (>2 classes of bDMARDs and/or tsDMARDs is exclusionary)

For axial spondyloarthritis:

* Moderate-to-severely active axSpA defined by BOTH of the following at Screening AND Day 1:

  1. BASDAI ≥4, AND
  2. Back pain ≥4 (from BASDAI Item 2)
* hsCRP greater than the ULN per the central laboratory at Screening
* Inadequate response (defined as signs and symptoms of persistently active disease, loss of response, or intolerance) to:

  1. 2 different NSAIDs given at the maximum tolerated dose for ≥4 weeks or intolerant to or has a contraindication to NSAID therapy; AND/OR
  2. ≤2 classes of bDMARD (anti-TNF or anti-IL-17)/tsDMARD at an approved dose for ≥12 weeks (>2 classes of bDMARDs/tsDMARDs is exclusionary)

For psoriatic arthritis:

* Screening and Day 1 TJC ≥3 out of 68 and SJC ≥3 out of 66 (dactylitis counts as 1 joint each)
* ≥1 active plaque psoriasis lesion and/or a documented history of psoriasis
* Inadequate response (defined as signs and symptoms of persistently active disease, loss of response, or intolerance) to:

  1. ≥1 NSAID treatment; AND
  2. ≥1 csDMARD treatment; AND/OR ≤2 classes of bDMARD/tsDMARD treatment (>2 classes of bDMARDs and/or tsDMARDs is exclusionary)

Exclusion Criteria:

* Inadequate response to >2 classes of bDMARDs/tsDMARDs
* Other autoimmune, rheumatologic, inflammatory diseases or pain-amplification syndromes that might confound the evaluations of efficacy of SPY072

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid Arthritis: Change from baseline in Disease Activity Score in 28 joints (c-reactive protein) (DAS-CRP) | Week 12
  The score is calculated based on the number of tender and swollen joints out of 28 assessed (TJC28 and SJC28), a measure of inflammation in the blood (c-reactive protein, CRP), and the subject's overall assessment of their health (patient global assessment). Scores range from 0-10. Higher scores indicate greater disease activity.
Axial Spondyloarthritis: Change from baseline in Ankylosing Spondylitis Disease Activity Score (ADAS) | Week 16
  The score combines 5 disease activity variables (back pain, duration of morning stiffness, patient global assessment of disease activity, peripheral pain/swelling and measure of inflammation) to measure disease activity. Lowest score is 0.6 and increases as disease worsens. Higher scores indicate greater disease activity.
Psoriatic Arthritis: Proportion of participants who achieve an American College of Rheumatology 20 Response Criteria (ACR20) response | Week 16
  The proportion of subjects who achieve at least 20% improvement in tender and swollen joint counts (TJC and SJC), and at least 20% improvement in 3 out of 5 other disease activity measures (patient global assessment, physician global assessment, patient pain assessment, health assessment questionnaire, and measure of inflammation) will be assessed.

SECONDARY OUTCOMES:
Rheumatoid Arthritis: Proportion of participants who achieve an ACR20 response | Week 12
  The proportion of subjects who achieve at least 20% improvement in tender and swollen joint counts, and at least 20% improvement in 3 out of 5 other disease activity measures will be assessed.
Axial Spondyloarthritis: Proportion of participants who achieve an Assessment of Spondyloarthritis International Society (40% improvement) (ASAS40) response | Week 16
  The proportion of subjects who achieve at least 40% improvement in at least 3 out of 4 key domains related to disease severity (patient global assessment of disease activity, back pain, physical function, inflammation) while not experiencing worsening in the remain domain will be assessed.
Psoriatic Arthritis: Change from baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) | Week 16
  The sum of 5 key disease variables (tender joint count, swollen joint count, patient pain assessment, patient global assessment of disease activity, and C-reactive protein) will be assessed. Scores range from 0.1 to 86. Higher score indicates higher disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: SKYWAY-RD Study Director, Study Director — Spyre Therapeutics
Locations (41):
- United States (13):
  - Site 113, Avondale, Arizona
  - Site 114, Chula Vista, California
  - Site 111, Covina, California
  - Site 108, Tujunga, California
  - Site 112, Upland, California
  - Site 107, Whittier, California
  - Site 109, Hialeah, Florida
  - Site 106, Ormond Beach, Florida
  - Site 110, Tampa, Florida
  - Site 104, Duncansville, Pennsylvania
  - Site 105, Corpus Christi, Texas
  - Site 103, Tomball, Texas
  - Site 102, Tomball, Texas
- Bulgaria (5):
  - Site 503, Lovech, Lovech
  - Site 502, Pleven, Pleven
  - Site 506, Plovdiv, Plovdiv
  - Site 505, Plovdiv, Plovdiv
  - Site 504, Varna, Varna
- Czechia (4):
  - Site 706, Hlučín, Hlučín
  - Site 702, Moravská Ostrava, Ostrava-město
  - Site 704, Pardubice, Pardubický kraj
  - Site 705, Prague, Praha, Hlavní Mesto
- Georgia (8):
  - Site 303, Tbilisi, K'alak'i T'bilisi
  - Site 304, Tbilisi, K'alak'i T'bilisi
  - Site 301, Tbilisi, K'alak'i T'bilisi
  - Site 307, Tbilisi, K'alak'i T'bilisi
  - Site 305, Tbilisi, K'alak'i T'bilisi
  - Site 308, Batumi
  - Site 302, Kutaisi
  - Site 306, Tbilisi
- Moldova (2):
  - Site 201, Chisinau
  - Site 202, Chisinau
- Poland (7):
  - Site 401, Krakow, Lesser Poland Voivodeship
  - Site 407, Nowa Sól, Lubusz Voivodeship
  - Site 403, Warsaw, Masovian Voivodeship
  - Site 402, Opole, Opole Voivodeship
  - Site 406, Gdynia, Pomeranian Voivodeship
  - Site 405, Warszawa, Pomeranian Voivodeship
  - Site 408, Elblag, Warmian-Masurian Voivodeship
- Spain (2):
  - Site 602, A Coruña, A Coruña
  - Site 604, Chiclana de la Frontera, Cadiz

IPD SHARING:
Plan to Share IPD: No